CLINICAL TRIAL: NCT05421494
Title: The Effectiveness of Online Revised Written Exposure Therapy for PTSD: Randomized Controlled Trials
Brief Title: The Effectiveness of Written Exposure Therapy for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yinyin Zang, PhD, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WET-R for PTSD
Record Dates: First submitted 2022-06-09; First posted 2022-06-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: PTSD; Subclinical PTSD
Keywords: PTSD; written exposure therapy; randomized controlled trial; online intervention; online psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- study2: WET-R (Experimental)
  Interventions: Behavioral: written exposure therapy-revised version
- study 2: MCC (Placebo Comparator)
  Interventions: Behavioral: minimal contact control
- study 1: WET (Experimental): Written Exposure Therapy (WET) is a manualized exposure-based therapy involving five sequential weekly individual sessions. Each session lasts approximately 40 minutes except the first, which is one hour. In the initial session, the therapist explains the treatment rationale and guides the participant to write about their traumatic experience uninterrupted for 30 minutes. Subsequent sessions start with a brief discussion about the previous session's writing, followed by another 30-minute writing session, concluding with a short check-in. There is no homework between sessions.
  Interventions: Behavioral: written exposure therapy-revised version
- study 1: WET+MBA (Experimental): WET + MBA combines the standard WET protocol with the addition of a mindfulness practice facilitated through a mobile app called "Now Meditation." This app is among the most downloaded mindfulness apps in China, used to help manage symptoms of insomnia commonly comorbid with PTSD. Participants are instructed to engage in daily mindfulness exercises according to the app's "7-Day Basic Meditation" program and continue practicing mindfulness throughout the duration of the therapy. This is intended to supplement the therapeutic effects of WET by providing tools to manage insomnia and potentially enhancing the therapeutic process by fostering greater mindfulness and relaxation.
  Interventions: Behavioral: written exposure therapy-revised version
- study 1: MCC (Placebo Comparator): MCC contains weekly phone calls from a study therapist to monitor their status and provide support as needed, without introducing any specific therapeutic interventions. These calls are brief, generally lasting between 10 to 15 minutes, and are strictly for the purpose of engagement and safety monitoring rather than therapeutic intervention.
  Interventions: Behavioral: minimal contact control

INTERVENTIONS:
Behavioral: written exposure therapy-revised version — WET-R is a manualized exposure-based therapy program consisting of 5-7 sequential individual sessions. The interval between every 2 consecutive sessions is 0-3 days. There will be 5-7 one to one online sessions in total (only one index trauma will be discussed), and 1-3 weeks to complete. Sessions are scheduled to last for 1 hour in the first session and 50 minutes in other sessions.
  Arms: study 1: WET; study 1: WET+MBA; study2: WET-R
Behavioral: minimal contact control — Participants assigned to MCC will be asked to not work with other therapists or seek additional treatment for trauma-related difficulties during the 3-week MCC period. They will be video-called once per week by a therapist to monitor their status and to provide support as needed. The calls will be limited to 10-15 minutes. MCC participants will also be given contact information to use in case of worsening symptoms or increasing distress.
  Arms: study 1: MCC; study 2: MCC

SUMMARY:
Study 1: The goal of this study is to use a pilot RCT to assess the effectiveness of Written Exposure Therapy (WET) and a mindfulness-based app (MBA) for managing PTSD and comorbid insomnia in China. The main questions it aims to answer are:

1. Does WET alone reduce PTSD symptoms in Chinese patients with PTSD and subthreshold PTSD?
2. Does the addition of MBA to WET lead to greater reductions in comorbid insomnia symptoms compared to WET alone?

45 participants will be allocated to MCC, WET, and WET+MBA on a 1:1:1 ratio. Researchers will compare WET alone and MCC to see if WET provides benefits in managing PTSD. Researchers will compare WET plus MBA and WET group to see if the integrated MBA treatment provides additional benefits in managing insomnia.

Study 2: The study aims to examine the effectiveness of the online revised written exposure therapy (WET-R) for PTSD and subclinical PTSD among Chinese adults with a randomized controlled trial. The study will recruit 90 participants, with 60 randomized to the online WET-R group, and 30 randomized to the minimal contact control (MCC) group. The WET-R intervention consists of 5-7 one to one sessions. The primary outcome PTSD Symptom Scale - Interview for DSM-5 (PSSI-5) will be administered on baseline, post-treatment, 1-month follow-up, 3-month follow-up, and 6-month follow-up assessments.

ELIGIBILITY:
Study 1:

Inclusion Criteria:

Adult male and female aged between 18-65 years old; A diagnosis of PTSD or subthreshold PTSD (PTSD Symptom Scale, Interview Version for DSM-5, PSSI-5); If currently taking psychotropic medication, taking a stable one for at least 4 weeks; A smartphone owner and no obstacle to the Now Meditation App; Scoring 12 or more on Insomnia Severity Index (ISI; the symptoms appear after the diagnosis of full/subthreshold PTSD).

Exclusion Criteria:

A diagnosis of bipolar disorder or psychotic disorder; Current substance dependence; Evidence of a moderate or severe traumatic brain injury (as determined by the obstacle to comprehending the baseline screening questionnaires); Serious suicidal ideation (as determined by the Scale for Suicidal Ideation); Other psychiatric disorders severe enough to warrant designation as the primary disorder; Taking psychotherapy for PTSD currently.

Study 2:

Inclusion Criteria:

1. Adult male and female (aged between 18-65 years old)
2. A diagnosis of PTSD or subclinical PTSD (PTSD Symptom Scale, Interview Version for DSM-5, PSSI-5), meeting the following criteria: Meeting full criteria for re-experiencing and at least 2 of 3 other symptom clusters (i.e., avoidance, negative cognitions, or hyperarousal)
3. If currently taking psychotropic medication, taking a stable one for at least 4 weeks
4. Having the ability to write and comprehend the writing guidelines

Exclusion Criteria:

1. A diagnosis of bipolar disorder or psychotic disorder
2. Current substance dependence
3. Evidence of a moderate or severe traumatic brain injury (as determined by the obstacle to comprehending the screening questionnaires)
4. Serious suicidal ideation (as determined by the MINI interview)
5. Taking psychotherapy for PTSD currently

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
study 2: Change from Baseline of PTSD Symptom Scale, Interview Version for DSM-5(PSSI-5) at Posttreatment | 3 weeks
  The PTSD Symptom Scale, Interview Version for DSM-5 (PSSI-5), a 24-item clinician-administered interview, will be used for PTSD diagnosis and measure PTSD symptom severity. The PSSI-5 rates the frequency and severity of PTSD symptoms in the past 4 weeks on a 5-point Likert scale from 0 (not at all) to 4 (very much). The PSSI-5 has demonstrated excellent reliability and validity but takes less time than the gold standard mostly used, the Clinician-Administered PTSD Scale for DSM-5 (CAPS5).
study 2: Change from Baseline of PTSD Symptom Scale, Interview Version for DSM-5(PSSI-5) at the First Follow-Up | 7 weeks
  The PTSD Symptom Scale, Interview Version for DSM-5 (PSSI-5), a 24-item clinician-administered interview, will be used for PTSD diagnosis and measure PTSD symptom severity. The PSSI-5 rates the frequency and severity of PTSD symptoms in the past 4 weeks on a 5-point Likert scale from 0 (not at all) to 4 (very much). The PSSI-5 has demonstrated excellent reliability and validity but takes less time than the gold standard mostly used, the Clinician-Administered PTSD Scale for DSM-5 (CAPS5).
study 2: Change from Baseline of PTSD Symptom Scale, Interview Version for DSM-5(PSSI-5) at the Second Follow-Up | 15 weeks
  The PTSD Symptom Scale, Interview Version for DSM-5 (PSSI-5), a 24-item clinician-administered interview, will be used for PTSD diagnosis and measure PTSD symptom severity. The PSSI-5 rates the frequency and severity of PTSD symptoms in the past 4 weeks on a 5-point Likert scale from 0 (not at all) to 4 (very much). The PSSI-5 has demonstrated excellent reliability and validity but takes less time than the gold standard mostly used, the Clinician-Administered PTSD Scale for DSM-5 (CAPS5).
study 2: Change from Baseline of PTSD Symptom Scale, Interview Version for DSM-5(PSSI-5) at the Third Follow-Up | 27 weeks
  The PTSD Symptom Scale, Interview Version for DSM-5 (PSSI-5), a 24-item clinician-administered interview, will be used for PTSD diagnosis and measure PTSD symptom severity. The PSSI-5 rates the frequency and severity of PTSD symptoms in the past 4 weeks on a 5-point Likert scale from 0 (not at all) to 4 (very much). The PSSI-5 has demonstrated excellent reliability and validity but takes less time than the gold standard mostly used, the Clinician-Administered PTSD Scale for DSM-5 (CAPS5).
study 1: PTSD symptom severity | Assessed at baseline, immediately post-treatment, and at 3-month follow-up periods.
  The reduction in PTSD symptoms will be measured using the PTSD Symptom Scale, Interview Version for DSM-5 (PSSI-5). This clinician-administered interview assesses the frequency and severity of PTSD symptoms using a 5-point Likert scale ranging from 0 (not at all) to 4 (very much).

SECONDARY OUTCOMES:
study 1: Insomnia Severity | Insomnia severity is assessed at baseline, weekly during the 5-week treatment period, and at the immediate post-treatment, and 3-month follow-up assessments.
  The reduction in the severity of insomnia symptoms will be assessed using the Insomnia Severity Index (ISI). This 7-item self-report measurement evaluates the severity of insomnia symptoms, the level of satisfaction with sleep, interference with daily functioning, noticeability of impairment attributed to sleep problems, and the level of distress caused by the sleep disturbance. Each item is rated on a 5-point scale, providing a comprehensive measure of insomnia severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided